CLINICAL TRIAL: NCT00846573
Title: Hyperpolarized Noble Gas MR Imaging for Pulmonary Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted prematurely as the PI was no longer an employee of UMass Medical School.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Mitchell Albert, Director of Advanced MRI Center, UMASS Medical Sch, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Docket # 12639
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: COPD; Cystic Fibrosis; Asthma; Healthy
Keywords: Helium; MRI; Hyperpolarized Helium; Hyperpolarized Noble Gas
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cystic Fibrosis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Asthmatic Participants (Experimental): This population is made up of only confirmed asthmatics. Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
  Interventions: Drug: Hyperpolarized Helium-3
- Healthy (Experimental): This population is made up of subjects who are considered clinically healthy. This means that there are no records of any chronic disorders or pulmonary history.
  Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
  Interventions: Drug: Hyperpolarized Helium-3
- COPD Patients (Experimental): This population is made up of only confirmed COPD patients. Diagnosis must be confirmed through their doctor prior to enrollment.
  Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
  Interventions: Drug: Hyperpolarized Helium-3
- Cystic Fibrosis Patients (Experimental): This population is made up entirely of confirmed cystic fibrosis patients. Diagnosis must be confirmed through their physician.
  Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
  Interventions: Drug: Hyperpolarized Helium-3

INTERVENTIONS:
Drug: Hyperpolarized Helium-3 — Patients will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
  Other Names: HP 3He

SUMMARY:
The purpose of this study is to test the efficacy of Hyperpolarized Helium-3 gas in MR imaging in COPD, asthmatics, CF and healthy volunteers.

DETAILED DESCRIPTION:
Current pulmonary imaging techniques are clinically regulated to machines that produce radiation. MR which does not produce radiation was not possible due to the low concentration of fluids in the open spaces of the lungs. With hyperpolarized noble gases we can now use the safe techniques of MR imaging to view the airways of the lungs, thus limiting human exposure to radiation. This technique has already been proven to be possible in human subjects but there is insufficient data show its efficacy in a clinical setting. This study is designed to image a variety of pulmonary disorders to better find possible clinical uses for hyperpolarized gas MRI.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female and are 5 years or older
* Consent/assent from the patient
* Have been diagnosed with a pulmonary disease such as COPD, Asthma, or cystic fibrosis. OR Healthy Individuals.
* Must be able to hold their breath for up to 15 seconds

Exclusion Criteria:

* Have any contraindications to an MR exam such as a pace-maker, metallic cardiac valves, magnetic material (i.e., surgical clips) implanted electronic infusion pumps or any other conditions that would preclude proximity to a strong magnetic field;
* Are undergoing the MR exam in an emergency situation
* Are pregnant or become pregnant at any point within the study time.
* People with psychiatric disorders will be excluded from the study.
* Are claustrophobic and can not tolerate the imaging.
* Uses supplemental oxygen

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Albert, Ph.D., Principal Investigator — UMASS Medical School
Locations (1):
- UMASS Medical School Advanced MRI Center United States, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began November 2008 and enrollment started January 2009. Recruitment continued until the study was terminated, April 2011. Participants were asthmatics, COPD patients, or CF patients as confirmed by their physician. Recruitment was completed from the UMass Memorial Medical Centre. Alternatively, healthy volunteers were also recruited.
Pre-assignment Details: Participants were excluded if their diagnosis of a lung condition could not be confirmed by medical records.
Groups:
- COPD: This population is made up of only confirmed COPD patients. Diagnosis must be confirmed through their doctor prior to enrollment.
  Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
- Asthma: This population is made up of only confirmed asthmatics. Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
- Cystic Fibrosis: This population is made up entirely of confirmed cystic fibrosis patients. Diagnosis must be confirmed through their physician.
  Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
Period: Overall Study
Arm/Group | COPD | Asthma | Cystic Fibrosis | Healthy
Started | 5 | 2 | 7 | 0
Completed | 5 | 2 | 7 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Asthma Patients: This population is made up of only confirmed asthmatics. Participants will inhale Hyperpolarized Helium-3: Participants will be required to breath in individual 1 liter bags of gas while in an MRI to produce lung images. These bags of gas are each made up of 333mL of Helium-3 gas and 667mL of Nitrogen. Three bags will be administered to acquire three different scans.
- Total: Total of all reporting groups
Arm/Group | COPD Patients | Asthma Patients | Cystic Fibrosis Patients | Total
Number analyzed (Participants) | 5 | 2 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 4 | 2 | 7 | 13
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (9.74) | 34.5 (14.85) | 27 (8.25) | 27.14 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 4 | 6
  Male | 3 | 2 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Hyperpolarized Helium-3 MR Images
Description: We have applied hyperpolarized 3He MR imaging to a range of subject with various disorders. We have developed our scanning techniques so as to acquire optimized images for each disorder.
Time Frame: 15 second breath-hold
Population: We recruited participants of each category until we were satisfied with the images we obtained.
Measure: Number; unit: participants
Arm/Group | COPD Patients | Asthma Patients | Cystic Fibrosis Patients
Number analyzed (Participants) | 5 | 2 | 7
participants | 5 | 2 | 7

ADVERSE EVENTS:
Arm/Group | COPD Patients | Asthma Patients | Cystic Fibrosis Patients
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less